CLINICAL TRIAL: NCT00727610
Title: Development of a Screening Strategy for Community-based Adverse Drug Related Events in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Patient Safety Institute (Other); Michael Smith Foundation for Health Research (Other); Vancouver Coastal Health (Other Government)
Responsible Party: Dr. Corinne M. Hohl/Scientist, University of British Columbia
Other Study IDs: H08-00510
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Adverse Drug Related Events
Keywords: Adverse drug event; harm; patient safety; clinical decision support; Adverse drug related event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Adverse Drug Related Events (ADREs) are a leading cause of Emergency Department (ED) visits in Canada. However emergency physicians recognize only half of all ADREs in patients presenting to the ED, missing opportunities to intervene. The objective of this study is to develop a screening strategy that identifies patients with ADREs. Our hypothesis is that the development of a user-friendly, reliable screening strategy for ADREs in patients presenting to the ED is feasible. We believe that this will lead to improved patient care.

DETAILED DESCRIPTION:
Background Between 9250 and 23,750 Canadians die each year because of preventable adverse events related to medical care. ADREs account for 50% of all preventable adverse events and cause up to 12% of ED visits. Unfortunately, emergency physicians recognize only half of all ADREs, missing crucial opportunities to intervene.

Objective The objective of this study is to derive a clinical decision rule that accurately stratifies patients presenting to the ED into risk categories for drug-related morbidity. This instrument will allow early identification of clinically significant ADREs allowing rational referral for medication optimization, treatment of ADREs and prevention of future events.

Hypothesis The development of a rapid, user-friendly reliable clinical decision rule for ADREs in patients presenting to the ED is feasible.

Methodology This prospective observational study will evaluate predictor variables (from the history, physical examination and laboratory tests) for ADREs in a representative sample of ED patients using standardized assessments by emergency nurses and physicians. Inter-rater agreement of predictor variables will be measured, and clinical pharmacists, blinded to the nursing and physician assessments, will use a standardized, validated algorithm to identify ADREs. Recursive partitioning and/or logistic regression analysis will be used to determine the optimal combination of predictor variables to detect the presence of an ADRE. We will report diagnostic test characteristics of the derived clinical decision rule. Validation of the clinical decision rule is planned in a future study.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19 years
* Reported having used at least one prescription or over-the-counter medication in the 2 weeks prior to presentation
* Speak English and/or translator available at the time of presentation.

Exclusion Criteria:

* Patients previously enrolled
* Patients transferred directly to an admitting service.
* Patients who leave prior to being seen or against medical advice.
* Patients returning to the ED for a scheduled revisit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the emergency departments of participating institutions who have used at least one prescription or over-the-counter medication in the 2 weeks prior to presentation.
Sampling Method: Probability Sample
Enrollment: 1588 (Estimated)
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Overall Officials: Corinne M. Hohl, Principal Investigator — University of British Columbia; Jeffrey R. Brubacher, Study Chair — University of British Columbia; Samuel B. Sheps, Study Director — University of British Columbia; Linda Dempster, Study Director — University of British Columbia; Garth Hunt, Study Director — University of British Columbia; Claude Stang, Study Director — University of British Columbia; Janet Joy, Study Director — University of British Columbia; Peter Loewen, Study Director — University of British Columbia; Matthew Wiens, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - Emergency Department, Vancouver General Hospital, Vancouver, British Columbia
  - Emergency Department, St Paul's Hospital, Vancouver, British Columbia